CLINICAL TRIAL: NCT04311008
Title: Turkish Version of Life Balance Inventory: Validity, Reliability and Cultural Adaptation
Brief Title: Turkish Life Balance Inventory
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İNAL, Trakya University, Hacettepe University
Other Study IDs: 2020/79
Record Dates: First submitted 2020-03-13; First posted 2020-03-17 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Version; Adaptation; Reliability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Turkish Version of Life Balance Inventory: Validity, Reliability and Cultural Adaptation.

DETAILED DESCRIPTION:
The Life Balance Inventory (Kathleen Matuska; 2012) is a measure for life balance. This study was planned for the purpose of carrying out Turkish Version of the Life Balance Inventory.

ELIGIBILITY:
Inclusion Criteria:

19-25 years old student at the Faculty of Health Sciences

-

Exclusion Criteria:

* not between age 19-25

Ages: 19 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: student at the Faculty of Health Sciences
Sampling Method: Probability Sample
Enrollment: 371 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2020-12-29 (Estimated); Study Completion 2020-12-29 (Estimated)

PRIMARY OUTCOMES:
Turkish Life Balance Inventory is Valid and Reliable | six months

CONTACTS AND LOCATIONS:
Overall Officials: Özgü İnal, Principal Investigator — Trakya University
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)